CLINICAL TRIAL: NCT05171712
Title: Portico and Navitor India Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10387
Record Dates: First submitted 2021-10-28; First posted 2021-12-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Failure; Aortic Insufficiency; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Analysis Population (Experimental): The analysis population will include patients considered at high or extreme surgical risk, who have met all inclusion criteria, have not met any exclusion criteria, have signed an Ethics Committee (EC) approved Informed Consent, and, at the minimum, the FlexNav delivery system entered his/her vasculature for an attempted Portico or Navitor Valve implant
  Interventions: Device: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement — Transcatheter Aortic Valve Replacement for the treatment of patients with severe aortic stenosis

SUMMARY:
The objective of this clinical trial is to collect data on procedural safety and device performance of the Portico and Navitor devices and FlexNav delivery system to treat patients with severe aortic stenosis in the Indian population.

DETAILED DESCRIPTION:
The objective of this Phase IV clinical trial is to characterize the procedural safety and device performance of the Portico valve, the Navitor Valve, the FlexNav delivery system and FlexNav or Navitor loading system to treat patients with severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation-related procedure.
2. Are >60 years of age in host country, have severe symptomatic (NYHA class ≥ II) aortic stenosis (AS), at high or extreme surgical risk and have been identified as a candidate for a Portico or Navitor valve implant.
3. Subjects must have a Society of Thoracic Surgeons (STS) score of ≥7% OR documented heart team agreement of high or extreme risk for surgical aortic valve replacement due to frailty or co-morbidities not captured by the STS score.

Exclusion Criteria:

1. Have tested positive for the Corona Virus Disease 2019 (COVID-19) virus at any time AND currently have residual signs or symptoms associated with the COVID-19 virus (eg. evidence of thrombosis, damaged/inflamed heart muscle, damaged/inflamed lung tissue, etc.)
2. Have sepsis, including active endocarditis
3. Have any evidence of left ventricular or atrial thrombus
4. Have vascular conditions (i.e. caliber, stenosis, tortuosity, or severe calcification) that make insertion and endovascular access to the aortic valve improbable
5. Have a non-calcified aortic annulus
6. Have congenital bicuspid or unicuspid leaflet configuration
7. Are unable to tolerate antiplatelet/anticoagulant therapy
8. Are pregnant at the time of signing informed consent
9. Are currently participating in a drug or device study that may impact this study (unless prior sponsor approval for co-enrollment is granted)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
VARC-2 and VARC-3 defined event rate of All cause mortality rate (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33
VARC-2 and VARC-3 defined event rate of Cardiovascular mortality rate (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Myocardial Infarction rate (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Stroke (including disabling and non-disabling, percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Bleeding (life-threatening, major, minor, percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Acute kidney injury (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Vascular access site and access-related complications (major and minor, percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Coronary obstruction (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Permanent pacemaker insertion (percent of subjects) at 30 days from the implant/index procedure | 30 days post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
Access Vessel Diameter (mm) during procedure | During procedure
  The access vessel diameter (mm) will be analyzed at index/implant procedure to define delivery profile characteristics
Sheath Utilization during procedure | During procedure
  The Sheath Utilization will be analyzed at index/implant procedure to define delivery profile characteristics (unit = percent using sheath)
Sheath Size during procedure | During procedure
  The Sheath Size will be analyzed at index/implant procedure to define delivery profile characteristics (unit = French (F))
Percentage of Subjects with Implant Success | During procedure
  Defined as absence of procedural mortality, correct positioning of a single Portico prosthetic heart valve into the proper anatomical location, no conversion to open surgery
Echocardiographic assessment of the mean gradient at 30 days compared to baseline for the subjects with Portico valve implanted | 30 days post index procedure
  Units=mmHg
Echocardiographic assessment of Effective Orifice Area (EOA) at 30 days compared to baseline for the subjects with Portico valve | 30 days post index procedure
  units = cm2
Echocardiographic assessment of Paravalvular Leak (PVL) per VARC-2 definitions at 30 days compared to baseline for the subjects with Portico valve implanted | 30 days post index procedure
  Reported as either none/trace, mild, moderate, or severe
VARC-2 and VARC-3 defined event rate of All-Cause Mortality (percent of subjects) beyond 30 days through 9 from the implant/index procedure | 9 months post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
VARC-2 and VARC-3 defined event rate of Stroke (including disabling and non-disabling, percent of subjects) beyond 30 days through 9 from the implant/index procedure | 9 months post index procedure
  The outcome measures will be defined for all VARC-2 and VARC-3 defined endpoints per the published VARC-2 and VARC-3 definitions:
  1. Kappetein et al. J Thorac Cardiovasc Surg: 2013;145:6-23.
  2. Genereux et al. European Heart Journal: 2021; 00, 1-33.
Clinical improvement from baseline to 30 days and baseline to 9-months for the subjects with Portico valve implanted assessed by New York Heart Association (NYHA) functional class | 30 days post index procedure
  Reported as the percent of subjects with improvement, worsening, or stable NYHA class from baseline to 30 days and from baseline to 9 months; NYHA Class will be measured as class I, II, III, or IV, symptoms are worsening from I to IV.
Clinical improvement from baseline to 30 days and baseline to 9-months for the subjects with Portico valve implanted assessed by Quality of Life (QoL) questionnaire (5-level EQ-5D version (EQ5D-5L)) | 9 months post index procedure
  Reported as the percent of subjects with improvement, worsening, or stable from baseline to 30 days and from baseline to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott
Locations (6):
- India (6):
  - Apollo Hospital, Chennai
  - Medanta-The Medicity, Gūrgaon
  - Rajasthan Hospital, Jaipur
  - Seth GS Medical College & KEM Hospital, Mumbai
  - Vardhman Mahavir Medical College & Safdarjung Hospital, New Delhi
  - Christian Medical College & Hospital, Vellore

IPD SHARING:
Plan to Share IPD: No